CLINICAL TRIAL: NCT06596096
Title: Risk Factors for Beta-lactam Target Non Attainment in Critically Ill Patients
Brief Title: Risk Factors for Beta-lactam Target Non Attainment in Critically Ill Patients BETALACTACRIT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Other Study IDs: CHSB-2022-08-P5-BETALACTACRIT
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Sepsis
Keywords: Beta-lactam; Underexposure; Risk factors; Intensive care unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Biological workup: hematological workup (CBC, platelets), blood urea, blood creatinine, urine urea, urine creatinine, blood gas, liver workup.
  * Plasma betalactamine determination (residual or steady-state).
  * Identification of bacteria responsible for infection inhibitory concentration value.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Beta-lactams agents are time-dependent antibiotics. Their bactericidal effects are associated with the time spent above the minimal inhibitory concentration (MIC) of the bacteria. In ICU patients, many pathophysiological changes may occur, which significantly alter beta-lactam pharmacokinetics (increasing in distribution volume, hypoalbuminemia or change in glomerular filtration rate…), leading to antibiotic underexposure, which may explain some treatment failures and risk of emergence of a multi-resistant bacteria.

Many guidelines advocate to reach a fixed target for the steady-state free plasma concentration of beta-lactam between 4 and 8 times of the MIC. However, clinical evidences supporting that septic patients in ICU would benefit from such optimization remain low and contradictory, and use of surrogate MICs based on critical breakpoints instead of actual MICs are significant limitations in the description of beta-lactam exposure among ICU patients with sepsis.

In this study, the investigators aim to indentify profiles of intensive care unit patients which are more likely to be associated with pharmacological failure (< 4 time the MIC of the bacteria). The investigators also aim to identify association between failure and poor clinical outcome.

DETAILED DESCRIPTION:
The duration of patient participation extends from the inclusion visit (D1), to discharge from intensive care; if the participant is still in intensive care at D90, the last visit with data collection will be at D90. The maximum duration of participation in the study will therefore be 3 months.

Taking into account 3 months of set-up, 1 year of recruitment, 3 months of participant follow-up, 3 months of data processing and 3 months of interpretation, 2 years will be sufficient to carry out this project.

ELIGIBILITY:
Inclusion Criteria:

* Participant over 18 years of age.
* Hospitalized in intensive care unit.
* Bacterial infection documented by culture.
* Treatment with beta-lactam for less than 48 hours.
* Person not objecting to participation in the study. If the particpant is unable to receive the information, it will be given to a relative and his or her non-opposition will be collected; the patient's non opposition will be sought and collected as soon as his or her condition permits.

Exclusion Criteria:

* Measurement of MIC of the bacterium in question impossible.
* Patients allergic to beta-lactam antibiotics.
* Patients with an estimated hospital stay of less than 3 days.
* Participants with "complex" infectious sites: central nervous system infection, osteoarticular infection, etc.
* Patients already included in the present study on the occasion of a previous beta-lactam administration.
* Adult patients under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care with sepsis.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Identify proportion of participant with betalactam underexposure in critically ill patients with sepsis and predictive parameters. | 25 months
  Under-exposure to beta-lactam antibiotics is defined as a plasma concentration below 4x the MIC of the identified bacterium. This concentration will be measured as residual in the case of discontinuous administration, or at equilibrium in the case of continuous administration. This criterion is assessed between 48 and 72 hours after the start of antibiotic therapy. Variables that will be assessed include age (in years), body mass index (in kg/m²), renal clearance (calculated with creatininemia, urinary creatininuria urinary volumeper day expressed in mL/min), SAPSII score (no unit), site of infection, modality of antibiotic administration (intermittent, continuous), time since first antibiotic injection (in hours), body temperature (in °C), SOFA score (no units), blood cell numeration (in cell/mL), coagulation parameters (in % of activity), protidemia (in g/L), lactates level (in mmol/L).

SECONDARY OUTCOMES:
Count the number of participants with poor clinical outcome and pharmacological failure (< 4 times the bacterial MIC). | 25 months
  The secondary objective is to establish the association between under-exposure to betalactam antibiotics in ICU participants and their clinical outcome. Pharmacological failure, defined as < 4 times the bacterial MIC, will be correlated with poor clinical outcome, up to and including death.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FILLATRE, Principal Investigator — CENTRE HOSPITALIER SAINT-BRIEUC PAIMPOL TREGUIER REANIMATION; Nicolas NESSELER, Study Chair — CHU RENNES REANIMATION CHIRURGIE THORACIQUE CARDIAQUE ET VASCULAIRE; Yoann LAUNEY, Study Chair — CHU RENNES REANIMATION CHIRURGICALE; Flora DELAMAIRE, Study Chair — CHU RENNES REANIMATION MEDICALE; Guillaume RIEUL, Study Chair — CH BRETAGNE ATLANTIQUE REANIMATION; Pierre BOUJU, Study Chair — ch bretagne sud atlantique REANIMATION; Aurélien FREROU, Principal Investigator — CH ST MALO REANIMATION
Locations (1):
- FILLATRE, Saint-Brieuc, France